CLINICAL TRIAL: NCT00950313
Title: Assessment of Response Rates and Yields for Two Tools for Early Detection of Non-diabetic Hyperglycaemia and Diabetes
Acronym: ATTEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 0132
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2009-07

CONDITIONS: Diabetes
Keywords: Diabetes; Screening; Risk; Self assessment
MeSH Terms: conditions — Diabetes Mellitus | interventions — Diagnostic Self Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self Assessment (Active Comparator): Patients are approached and asked to complete a risk score that will determine their current risk of diabetes and the likelihood of requiring further testing.
  Interventions: Other: Self Assessment
- Electronic risk score (Active Comparator): Patients diabetes riks is determined based on their data held on practice systems. Patients are then invited for further testing based on this score.
  Interventions: Other: Electronic risk score

INTERVENTIONS:
Other: Self Assessment — Self assessment used to determine current risk of diabetes and likelihood of requiring further testing
  Arms: Self Assessment
Other: Electronic risk score — Patients current risk of diabetes is determined by a electronic risk algorithm. They are then invited to attend fof further testing.
  Arms: Electronic risk score

SUMMARY:
The purpose of this study is to establish the most effective method of increasing attendance to screening of type 2 Diabetes within a primary care setting within the backdrop of the NHS Health Check programme.

DETAILED DESCRIPTION:
The University Hospitals of Leicester and The University of Leicester have developed a self-assessment risk score and a practice data risk score that can be used in a variety of setting to detect undiagnosed diabetes and impaired glucose regulation. This is done to establish a simple and effective 1st stage screen to identify those people at risk of diabetes and engage the public to increase the number of high risk individuals attending screening invitations but reducing the overall number of oral glucose tolerance tests. This study aims to test in a pragmatic way the use of such tools in a primary care setting administered by primary care staff as part of the NHS Health Check programme.

ELIGIBILITY:
Inclusion Criteria:

* 40-75 years old (30 -75 years old if South Asian origin)

Exclusion Criteria:

* Current diagnosis of diabetes
* Terminal illness or mental incapacity

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Increase in response rates to invitation to 2nd stage blood test | 12 months

SECONDARY OUTCOMES:
Increase in yield of OGTT positive results through filtering of high risk participants that pass 1st and 2nd stage screens | 12

CONTACTS AND LOCATIONS:
Overall Officials: Kamlesh Khunti, MD, Principal Investigator — University of Leicester
Locations (1):
- Leicester City PCT, Leicester, Leicestershire, United Kingdom